CLINICAL TRIAL: NCT04279366
Title: Evaluation and Validation of Biological Age as Health Technology
Brief Title: Biological Age Applied at Ubberup
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Jørn Wulff Helge, Proffesor Jørn Wulff Helge, University of Copenhagen
Other Study IDs: UbberupBioAge
Record Dates: First submitted 2020-02-18; First posted 2020-02-21 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Healthy Aging; Lifestyle Risk Reduction
Keywords: Individualised Health; Prediction; Risk Assessment
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Weeks
Biospecimen Retention: Samples With DNA — Blood sample will be drawn from a vein in the elbow
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Winter course: The recruited particpants attending the winter course
  Interventions: Behavioral: Lifestyle intervention
- Fall course: The recruited particpants attending the winter course
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — The 14 week courses takes place at a Danish folk high school (Ubberup), specialized in lifestyle interventions targeting a 10% weight loss. Adult individuals with obesity sign up for the course. They stay at the School for the whole course period and the total cost amounts to 300-400 Euros per week plus loss of income.

SUMMARY:
In a previous study the investigators have developed a novel biological age model. Assessing biological age is the assessment of the present health status and functional capacity/physiological reserve of that person in comparison with people of the same age and sex.

The aim of this study is to investigate the utility and validity of this novel biological age model designed for health promotion in real world conditions.

DETAILED DESCRIPTION:
Study design: This is a longitudinal study, where biological age assessment is conducted in the first and final week of an 11-14 week lifestyle intervention course. These courses take place at a Danish folk high school (Ubberup), which is specialized in performing intensive lifestyle interventions targeting a 10% weight loss. The intention is to include 80 adult men and women.

Data collection: This will take place at the facilities at Ubberup folk high school, participants being overnight fasted and without having exercised for the previous 24 hours. All analysis will be performed in investigators lab (Xlab) at the Department of Biomedical Sciences, Copenhagen University. When all samples are analysed Biological age will be calculated for each particpant.

ELIGIBILITY:
Inclusion Criteria:

* Participation in a long course at Ubberup folk high school (12-15 weeks)
* Age between 18-65 years

Exclusion Criteria:

* Previous or current cardiovascular disease
* Pregnancy
* Conditions that prevents from performing a cycle and/or strength tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adults participating and finishing the 12-14 week intensive lifestyle intervention at Ubberup folk high school.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Change in biological age | week1 and week 14
  a composite score predicting risk of lifestyle related diseases

SECONDARY OUTCOMES:
Change in cardiorespiratory capacity | week 1 and week 14
  VO2max maximal oxygen consumption (ml/min/kg
Change in strength | week 1 and week 14
  Hand grip, isometric quadriceps and biceps strength (Nm)
Change in Sit to Stand test | week 1 and week 14
  Rise and sit from a chair as many times as possible during 1 minute (number og rises)
Change in Central obesity | week 1 and week 14
  Waist to hip ratio is measured by dividing waist circumference with hip circumference in cm.
Change in body weight | week 1 and week 14
  measured in kilograms
Change in body composition | week 1 and week 14
  BMI (kg/m2) is calculated
Change in fat mass | week 1 and week 14
  fat mass(g) is assessed by bioimpedance
Change in fat percentage | week 1 and week 14
  Fat%, is assessed by bioimpedance
Change in muscle mass | week 1 and week 14
  muscle mass(g) is assessed by bioimpedance
Change in lipid profile | week 1 and week 14
  HighDensityLipoprotein (mmol/L), LowDensityLipoprofile (mmol/L), TriGlycerides (mmol/L), FreeFattyAcids (mmol/L) and Glycerol (mmol/L) is measured in a blood sample.
Change in Inflammatory profile | week 1 and week 14
  C-reactive protein mg/L, soluble urokinase plasminogen activating receptor ng/ml, InterLeukin 6 and 8 (pg/mL), tumor necrosis factor (pg/mL), Leptin and Adiponectin (ng/ml) is analysed from blood samples
Change in Blood glucose | week 1 and week 14
  HbA1c and fasting glucose (mmol/L) measured from blood sample
Change in Respirometry | week 1 and week 14
  forced vital capacity and forced expiratory volume at one second(L)
Change in Blood Pressure | week 1 and week 14
  Systolic and Diastolic blood pressure (mmHg)
Change in Advanced glycation endproducts | week 1 and week 14
  Levels of glycated protein and lipids as a result of exposure of excess sugars advanced glycation endproducts (AGE) measured in the skin
Change in Hormones | Week 1 and week 14
  Insulin

OTHER OUTCOMES:
Change in Metabolic Syndrome occurrence | week 1 and week 14
  A cluster of 5 risk factors predicting risk of CVD and T2D
Change in Framingham Risk Score | week 1 and week 14
  A composite score predicting 10 years risk of future CVD

CONTACTS AND LOCATIONS:
Overall Officials: Jørn W Helge, PhD, Principal Investigator — University of Copenhagen
Locations (2):
- Denmark (2):
  - Ubberup High School, Kalundborg, Danmark
  - Xlab, Faculty of Health and Medical Sciences, University of Copenhagen, Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Husted KLS, Fogelstrom M, Hulst P, Brink-Kjaer A, Henneberg KA, Sorensen HBD, Dela F, Helge JW. A Biological Age Model Designed for Health Promotion Interventions: Protocol for an Interdisciplinary Study for Model Development. JMIR Res Protoc. 2020 Oct 26;9(10):e19209. doi: 10.2196/19209. PMID 33104001